CLINICAL TRIAL: NCT02541162
Title: Cancer and Sexual Health : Early Information and Sexual Satisfaction of Couples in Oncology
Acronym: COUPLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was suspended because the oncology service decided to adopt the procedure in routine
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A00443-44
Record Dates: First submitted 2015-08-21; First posted 2015-09-04 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INFORMED (Experimental): Interventional Group (I): Couples enrolled during the diagnosis will receive written information as usual about the disease and in addition they benefit special oral interviews and written information about experiences of their sexuality during the illness.The document used for the interventional group is "Sexuality and Cancer" and will be given to couples. (intervention: Oral information and interviews about sexuality and self experience during the disease). Qualitative analysis will be provided by a psychologist
  Interventions: Behavioral: Oral information and interviews
- ORDINARY USE (No Intervention): Non-interventional Group (NI): Couples enrolled during the diagnosis will only receive written information about their experience of disease . The document used fot the non interventional group is "Live during and after cancer"and will be given to couples. Qualitative analysis will be provided by a psychologist

INTERVENTIONS:
Behavioral: Oral information and interviews — interviews about sexuality and self experience during the disease
  Arms: INFORMED

SUMMARY:
In a perspective of improvement of the global care of the patients, investigators wish to estimate, within the oncology department of Paris Saint Joseph Hospital, the impact of a clear, written and oral information, on the sexual satisfaction of the couples during treatments.

Further to this study, the project will be to train and to sensitize the medical staff, or still to develop new activities to meet the needs better of patients and of partners.

DETAILED DESCRIPTION:
To answer the objective, investigators set up a longitudinal study of a maximum duration of 18 months to recruit a minimum of 60 couples distributed in two groups:

The inclusion in the study will be made in two phases:

* The couples of the non-interventional group (NI) will be recruited at first to avoid the possibility to of sharing information between patients on their care. Indeed, it is about a comparative study and it is necessary that the couples of the NI group do not know about information proposed to the group I, at the risk of cancelling the effect of the information.
* The couples of the interventional group (I) will so be recruited during the last phase of the study of the NI group, that is approximately 6 months after the beginning of the study.

The choice of the minimal size of participants' sample is stretched out by the necessity of a minimum number of 30 participants by group to make relevant statistical analyses.

Once the information were given to the patients and to the partners, according to the group in which they are included, the participants will perform individually same sets of validated questionnaires at three different point times:

* initial visit: at the inclusion
* intermediate visit: 2 months after the inclusion
* final visit: 6 months after the inclusion

The Questionnaires will be manage through a local statistical analysis. The set of analyses will be led thanks to the statistical software SPSS. Descriptive analyses of the data, the correlations between the variables of the study and finally the tests of comparison will be perform to have an objective assessment criterion for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients and partners declaring itself in couple or having a shared private life;
* Patients diagnosed by an initial cancer, the prognosis for survival of which at the time of the diagnosis is upper to one year;
* Patients and partners of more than 18 years old, mastering the French language, and in measure to give their informed consent

Exclusion Criteria:

* Patients having been diagnosed and/or treated for another cancer;
* Patients and partners having a psychiatric disorder (confusional syndrome, psychotic disorders, disrupted reality perception)
* Patients and partners protected by the law, according to articles L.1121-5 to L.1121-8 of the Public health code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06-11 (Actual); Primary Completion 2015-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Quality Life (QLQ C30) due to a specific information about the sexuality on the sexual satisfaction of the couples, assessed | Participants will be followed during 6 months
  3 times points: Randomization (Day 1), 2 months and 6 months post-inclusion

SECONDARY OUTCOMES:
Change from baseline in Sexual Satisfaction Score (ESS) due to a specific information about the sexuality on the sexual satisfaction of the couples, assessed | Participants will be followed during 6 months
  3 times points: Randomization (Day 1), 2 months and 6 months post-inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Helene Beaussier, Pharm D, Study Director — CRC - GHPSJ
Locations (2):
- France (2):
  - hopital Saint Joseph, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided